CLINICAL TRIAL: NCT03073941
Title: A Multicenter Prospective Randomized Control Study on Persona Total Knee System vs NexGen Total Knee System in Total Knee Arthroplasty
Brief Title: A Multicenter Prospective Randomized Control Study on Persona Total Knee System vs NexGen
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K.CR.I.EU.15.13
Record Dates: First submitted 2017-01-17; First posted 2017-03-08 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee arthroplasty; Knee function; Total knee replacement; Persona total knee system; NexGen total knee system
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Persona CR (Active Comparator): Patients who received a Persona CR total knee implant
  Interventions: Device: Persona total knee system
- NexGen CR (Active Comparator): Patients who received a NexGen CR total knee implant
  Interventions: Device: Nexgen total knee system

INTERVENTIONS:
Device: Persona total knee system — 314 participants with knee osteoarthritis set to receive primary total knee arthroplasty will receive either Persona knee or the Nexgen
  Other Names: Zimmer Biomet Persona total knee system
  Arms: Persona CR
Device: Nexgen total knee system — 314 participants with knee osteoarthritis set to receive primary total knee arthroplasty will receive either Persona knee or the Nexgen
  Other Names: Zimmer Biomet Nexgen total knee system
  Arms: NexGen CR

SUMMARY:
A multicenter, prospective randomized controlled trial comparing the Persona knee system to the Nexgen knee system in total knee arthroplasty.

DETAILED DESCRIPTION:
Knee replacement is an established treatment for late stage osteoarthritis (OA) of the knee. There is an increasing demand for joint replacement in a younger population. Due to the changing demographics of joint replacement, the population of younger patients are seeking options that not only correct their disease or deformity, but do not limit them in activity. Studies have shown that modern implant designs can potentially improve outcome. Therefore new implants are introduced to the marked with the theoretical benefit of improved implant survival and superior patient reported outcomes. Within Total knee arthroplasty, design changes are introduced in an attempt to improve knee kinematics, functionality and outcome, but those potential improvements need to be evaluated.

The NexGen Total Knee System is a knee replacement system with well a documented performance and has been the device of choice in many institutions. Recently, Zimmer-Biomet have introduced Persona Total Knee system with design changes that include asymmetric tibia plate, increased medial pivoting and more extensive choices in respect to poly thickness, all with the purpose to improve balancing, stability and longevity. Such design changes and proposed benefits need to be evaluated in a prospective clinical trial, with focus on patient safety, satisfaction and implant durability.

The aim is to evaluate intra-operative and postop complications, long-term survivorship and patient reported outcome measures following primary total knee replacement using Persona Cruciate Retaining (CR) total Knee system compared to NexGen Cruciate Retaining (CR) total Knee System.

This project is carried out as a 2-arm randomized controlled single-blinded trial. A total of 314 participants are to be included at 6 centers in Denmark. Participants are seen on an outpatient basis at 3 months and 1 and 2 years postoperatively. After 2-year follow-up the patients will be followed for survivorship through the Danish Knee Arthroplasty Registry.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological osteoarthritis of the knee set to receive a primary unilateral total knee replacement
* >18 years of age
* Participants must be able to speak and understand Danish
* Participants must be able to give informed consent and be cognitively intact
* Participants must be able to complete all post-operative controls
* Participants must not have severe comorbidities, American Society of Anesthesiologists (ASA) score ≤ 3
* Clinically suitable to receive a CR implant (no severe deformity and/or ligament instability)

Exclusion Criteria:

* Terminal illness
* Revision knee replacement surgery
* Rheumatoid Arthritis (RA)
* Traumatic etiology
* Prior surgery on the affected knee that includes osteosynthesis, Anterior cruciate ligament (ACL) and/or Posterior cruciate ligament (PCL) and/or collateral ligament surgery. Arthroscopy with meniscectomy / cartilage surgery / house cleaning is allowed.
* Altered pain perception and / or neurologic affection due to diabetes or other disorders.
* Patients will be excluded intraoperative if CR implant is not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2031-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, Professor, Principal Investigator — Hvidovre University Hospital
Locations (5):
- Denmark (5):
  - Dept. of Orthopaedic Surgery, Farsø Sygehus, Ålborg Universitetshospital, Aalborg
  - Copenhagen University hospital, Gentofte, Copenhagen
  - Hvidovre hospital, Copenhagen
  - Dept. of Orthopaedic Surgery, Næstved Sygehus, Næstved
  - Dept. of Orthopaedic Surgery, Vejle Sygehus, Sygehus Lillebælt, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortensen KRL, Ingelsrud LH, Odgaard A, Kappel A, Varnum C, Schroder H, Gromov K, Troelsen A. Patient-reported outcomes and complications of a new-generation total knee system: a randomized controlled trial. Acta Orthop. 2025 Feb 25;96:195-202. doi: 10.2340/17453674.2025.43004. PMID 39998994

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 patients not assigned to any group: 5 rescinded consent before surgery, 13 recorded as lost to follow-up for other reasons
Period: Overall Study
Arm/Group | Persona CR | NexGen CR
Started | 157 | 157
Completed | 146 | 145
Not Completed | 11 | 12
Not completed — Received non-study device intraoperatively | 0 | 2
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 5 | 4
Not completed — Adverse Event | 4 | 2
Not completed — Met an exclusion criterion | 0 | 1

BASELINE CHARACTERISTICS:
Population: 157 patients were enrolled and randomized to each group, but 3 cases were excluded intraoperatively: 2 in the NexGen group and 1 in the Persona group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Persona CR | NexGen CR | Total
Number analyzed (Participants) | 156 | 155 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.2) | 67.7 (9.0) | 67.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 90 | 189
  Male | 57 | 65 | 122
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 156 | 155 | 311

OUTCOME MEASURES:

1. Primary Outcome: Oxford Knee Score
Description: The OKS is a patient-reported outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following TKA. The OKS consists of twelve questions covering function and pain associated with the knee. To calculate the total score, each question is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: 157 patients were enrolled and randomized to each group, but 3 cases were excluded intraoperatively: 2 in the NexGen group and 1 in the Persona group. Additionally, some data points are missing due to missed follow-up visits or incomplete form completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
score on a scale
  Preoperative: number analyzed (Participants) | 156 | 154
  Preoperative | 22.1 (6.7) | 22.2 (6.5)
  3 months: number analyzed (Participants) | 154 | 151
  3 months | 33.5 (7.8) | 32.9 (7.9)
  1 year: number analyzed (Participants) | 149 | 151
  1 year | 39.5 (7.7) | 38.6 (7.6)
  2 years: number analyzed (Participants) | 142 | 147
  2 years | 40.7 (7.3) | 40.8 (6.6)
Statistical Analysis 1: Comparison: Persona CR vs NexGen CR; Test type: Non-Inferiority — A non-Inferiority analysis was performed once the 1 year OKS of the first 216 patients were collected. A one-sided T-test, 90% power, SD=10 and with a non-inferiority margin of 4 OKS was used and the analysis was based on the difference of average OKS between Persona and NexGen 1 year postoperatively; p < 0.05, t-test, 1 sided; 90% power, SD=10 and with a non-inferiority margin of 4 OKS

2. Secondary Outcome: Oxford Knee Score - Activity & Participation Questionnaire (APQ)
Description: The OKS-APQ is an 8 item questionnaire with each question scored from 0 (worst outcome) to 4 (best outcome). The resulting score is then summed and converted to a score ranging from 0 (worst possible score) to a maximum of 100 (best possible score).
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
score on a scale
  Preoperative: number analyzed (Participants) | 156 | 154
  Preoperative | 16.4 (19.7) | 15.2 (19.4)
  3 months: number analyzed (Participants) | 154 | 151
  3 months | 50.0 (30.8) | 49.3 (30.5)
  1 year: number analyzed (Participants) | 149 | 151
  1 year | 71.4 (30.4) | 64.3 (31.9)
  2 years: number analyzed (Participants) | 142 | 147
  2 years | 70.5 (31.2) | 69.4 (31.0)

3. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The FJS-12 is a patient-reported outcome questionnaire that was developed to specifically assess the patient's level of awareness of the joint during daily activities. The FJS consists of twelve questions covering function and pain associated with the knee. For each question, there is a choice of five answers between never (0), almost never (1), seldom (2), sometimes (3) and mostly (4). All scores are summed up and divided by the number of completed items. This value is then multiplied by 25 and thereafter subtracted from 100. An outcome score of 100 (highest possible score) indicates the lowest level of joint awareness, while a total score of 0 indicates the highest level of joint awareness.
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
score on a scale
  Preoperative: number analyzed (Participants) | 156 | 154
  Preoperative | 14.3 (13.7) | 14.1 (13.4)
  3 months: number analyzed (Participants) | 154 | 151
  3 months | 42.8 (27.8) | 42.6 (26.0)
  1 year: number analyzed (Participants) | 149 | 151
  1 year | 60.3 (27.8) | 56.2 (29.2)
  2 years: number analyzed (Participants) | 142 | 147
  2 years | 65.0 (29.0) | 64.3 (27.0)

4. Secondary Outcome: Patient Satisfaction and Anchoring Questions - Question 1
Description: Patients were asked to answer the following satisfaction/anchoring question: "How are your knee problems now, compared to prior to your operation?"
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
Participants
  3 months: number analyzed (Participants) | 154 | 151
  3 months: Better, an important improvement | 109 | 99
  3 months: Somewhat better, but enough to be an important improvement | 31 | 33
  3 months: Very small change, not enough to be an important improvement | 6 | 7
  3 months: About the same | 3 | 4
  3 months: Very small change, not enough to be an important worsening | 2 | 4
  3 months: Somewhat worse, but enough to be an important worsening | 2 | 3
  3 months: Worse, an important worsening | 0 | 0
  3 months: Better, an important improvement + About the same | 1 | 0
  3 months: Very small change,not enough to be an important worsening + Somewhat worse | 0 | 1
  1 year: number analyzed (Participants) | 149 | 151
  1 year: Better, an important improvement | 123 | 111
  1 year: Somewhat better, but enough to be an important improvement | 16 | 29
  1 year: Very small change, not enough to be an important improvement | 6 | 2
  1 year: About the same | 0 | 1
  1 year: Very small change, not enough to be an important worsening | 2 | 0
  1 year: Somewhat worse, but enough to be an important worsening | 1 | 5
  1 year: Worse, an important worsening | 1 | 3
  1 year: Better, an important improvement + About the same | 0 | 0
  1 year: Very small change,not enough to be an important worsening + Somewhat worse | 0 | 0
  2 years: number analyzed (Participants) | 142 | 147
  2 years: Better, an important improvement | 118 | 123
  2 years: Somewhat better, but enough to be an important improvement | 18 | 19
  2 years: Very small change, not enough to be an important improvement | 3 | 2
  2 years: About the same | 1 | 0
  2 years: Very small change, not enough to be an important worsening | 1 | 1
  2 years: Somewhat worse, but enough to be an important worsening | 1 | 1
  2 years: Worse, an important worsening | 0 | 1
  2 years: Better, an important improvement + About the same | 0 | 0
  2 years: Very small change,not enough to be an important worsening + Somewhat worse | 0 | 0

5. Secondary Outcome: Patient Satisfaction and Anchoring Questions - Question 2
Description: Patients were asked to answer the following satisfaction/anchoring question: "Taking into account all the activities you have during your daily life, your level of pain and functional impairment, do you consider that your current state is satisfactory?"
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
Participants
  3 months: number analyzed (Participants) | 154 | 151
  3 months: Yes | 122 | 119
  3 months: No | 32 | 32
  1 year: number analyzed (Participants) | 149 | 151
  1 year: Yes | 127 | 132
  1 year: No | 22 | 19
  2 years: number analyzed (Participants) | 142 | 147
  2 years: Yes | 130 | 137
  2 years: No | 12 | 10

6. Secondary Outcome: Patient Satisfaction and Anchoring Questions - Question 3
Description: Patients were asked to answer the following satisfaction/anchoring question: "If you answered No, i.e. not satisfied to the result would you consider your current state as being so unsatisfactory that you think the treatment has failed?"
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 32 | 32
Participants
  3 months: Yes | 5 | 1
  3 months: No | 27 | 29
  3 months: No answer provided | 0 | 2
  1 year: number analyzed (Participants) | 22 | 19
  1 year: Yes | 4 | 8
  1 year: No | 18 | 11
  1 year: No answer provided | 0 | 0
  2 years: number analyzed (Participants) | 12 | 10
  2 years: Yes | 4 | 4
  2 years: No | 8 | 5
  2 years: No answer provided | 0 | 1

7. Secondary Outcome: Patient Satisfaction and Anchoring Questions - Question 4
Description: Patients were asked to answer the following satisfaction/anchoring question: "Would you have your knee operated again?"
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
Participants
  3 months: number analyzed (Participants) | 154 | 151
  3 months: Yes, definitely | 112 | 116
  3 months: Maybe, don't know | 32 | 27
  3 months: No | 10 | 8
  1 year: number analyzed (Participants) | 149 | 151
  1 year: Yes, definitely | 121 | 119
  1 year: Maybe, don't know | 25 | 25
  1 year: No | 3 | 7
  2 years: number analyzed (Participants) | 142 | 147
  2 years: Yes, definitely | 114 | 114
  2 years: Maybe, don't know | 22 | 23
  2 years: No | 6 | 10

8. Secondary Outcome: EuroQol 5D (EQ-5D) Score
Description: The EQ-5D is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, self-care, daily/usual activities, pain/discomfort and anxiety/depression.
  For EQ-5D-3L, each question can be answered in three ways, indicating no, moderate, or extreme pain. In the derived EQ-5D-3L score, the highest score is 1 and the lowest score is -0.59; negative numbers correspond to a self-assessed health state worse than being dead.
Time Frame: 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
score on a scale
  Preoperative: number analyzed (Participants) | 156 | 154
  Preoperative | 0.500 (0.272) | 0.516 (0.272)
  3 months: number analyzed (Participants) | 154 | 151
  3 months | 0.765 (0.190) | 0.778 (0.173)
  1 year: number analyzed (Participants) | 149 | 151
  1 year | 0.840 (0.201) | 0.840 (0.173)
  2 years: number analyzed (Participants) | 142 | 147
  2 years | 0.868 (0.187) | 0.866 (0.197)

9. Secondary Outcome: Radiolucency / Osteolysis
Description: All X-rays were sent to an independent radiographer. Postoperative lucency was determined as presence of radiolucent intervals at the cement-bone interface. Femoral lucency and tibial lucency are reported separately.
Time Frame: Immediate postoperative and 3 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Persona CR | NexGen CR
Number analyzed (Participants) | 156 | 155
Participants
  Immediate postoperative : Tibial lucency | 0 | 0
  Immediate postoperative : Femoral lucency | 1 | 2
  3 months : Tibial lucency: number analyzed (Participants) | 156 | 151
  3 months : Tibial lucency | 3 | 9
  3 months : Femoral lucency: number analyzed (Participants) | 156 | 152
  3 months : Femoral lucency | 7 | 9
  1 year : Tibial lucency: number analyzed (Participants) | 150 | 147
  1 year : Tibial lucency | 6 | 16
  1 year : Femoral lucency: number analyzed (Participants) | 150 | 147
  1 year : Femoral lucency | 14 | 22
  2 years : Tibial lucency: number analyzed (Participants) | 144 | 142
  2 years : Tibial lucency | 14 | 16
  2 years : Femoral lucency: number analyzed (Participants) | 144 | 142
  2 years : Femoral lucency | 21 | 20

10. Secondary Outcome: Long-term Survivorship
Description: Registry data at 5, 7 and 10 years postoperatively.
Time Frame: 5, 7 and 10 years postoperatively.
Reporting Status: Not Posted, anticipated posting 2031-12

ADVERSE EVENTS:
Time Frame: From study start up to 2 years post-operatively
Description: Adverse events have been documented continuously by checking with the study patients at every follow-up visit.
Groups:
- Persona CR: Patients who received a Persona CR total knee implant, excluding the 1 case excluded intraoperatively.
- NexGen CR: Patients who received a NexGen CR total knee implant, excluding the 2 cases excluded intraoperatively.
Arm/Group | Persona CR | NexGen CR
All-Cause Mortality (participants affected / at risk) | 1/156 | 0/155
Serious Adverse Events (participants affected / at risk) | 23/156 | 28/155
Other Adverse Events (participants affected / at risk) | 16/156 | 20/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona CR (N=156) | NexGen CR (N=155)
Arythmia (Cardiac disorders) | 0 (0) | 4 (4)
Congestive Hearth Failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis (Endocrine disorders) | 0 (0) | 1 (1)
Infection (non-knee) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gallstone + Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Shoulder Fracture Due to Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Knee Pain Due to Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Patella Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Patella Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trochanteric Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Nerve Injury (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Shortness of Breath/Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bowel Rupture (Surgical and medical procedures) | 0 (0) | 1 (1)
Contralateral Knee Replacement (Surgical and medical procedures) | 3 (3) | 5 (5)
Foot Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric Bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Spinal Stenosis (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cerebral Aneurysma (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemia + Influenza (Infections and infestations) | 0 (0) | 1 (1)
Revision Contralateral Knee (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tibial Base Plate Loosening (Surgical and medical procedures) | 0 (0) | 1 (1) — Revision surgery performed, all components revised
Infection (knee) (Surgical and medical procedures) | 0 (0) | 1 (1) — Revision surgery performed, all components revised
Dislocated Liner (Surgical and medical procedures) | 1 (1) | 0 (0) — Revision surgery performed, only liner revised
Knee Instability (Surgical and medical procedures) | 2 (2) | 0 (0) — Revision surgery performed, only liner revised
Flexion Contracture (Surgical and medical procedures) | 1 (1) | 0 (0) — Revision surgery performed, all components revised
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona CR (N=156) | NexGen CR (N=155)
Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Contralateral Knee Replacement (Surgical and medical procedures) | 0 (0) | 4 (4) — Planned hospitalization for a pre-existing condition (bilateral osteoarthritis)
Delayed Wound Healing (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Effusion (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — No hospitalization required
Flexion Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) — No hospitalization required
Knee Pain Due to Fall (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — No hospitalization required
Knee Swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Knee Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — No hospitalization required

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03073941/Prot_SAP_000.pdf